CLINICAL TRIAL: NCT05316636
Title: Randomized Clinical Trial on the Effect of Intermittent Vibrational Force Application During Orthodontic Treatment With Aligners on RANKL and OPG Concentrations in Crevicular Fluid
Brief Title: Intermittent Vibrational Force During Orthodontic Treatment With Aligners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Spanish Society of Orthodontics (SEDO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.P. - C.I. 15/313
Record Dates: First submitted 2022-03-21; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Orthodontic Tooth Movement; Gingival Crevicular Fluid; Biomarkers
Keywords: Vibration forces
MeSH Terms: interventions — Orthodontics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Vibrational forces from onset of treatment, from weeks 0-6; then, no vibrational forces during the rest of the treatment
  Interventions: Device: Vibrational forces; Procedure: Orthodontic treatment with clear aligners
- Group B (Experimental): From weeks 0-6, no vibrational forces. Vibrational forces starting at 6 weeks after treatment onset and applied for 6 weeks until week 12
  Interventions: Device: Vibrational forces; Procedure: Orthodontic treatment with clear aligners
- Group C (Active Comparator): Control, no vibrational forces
  Interventions: Procedure: Orthodontic treatment with clear aligners

INTERVENTIONS:
Device: Vibrational forces
  Arms: Group A; Group B
Procedure: Orthodontic treatment with clear aligners

SUMMARY:
This three-arm cross-over randomized clinical trial (allocation ratio of 1:1:1) will aim to explore whether the application of intermittent vibratory forces modify RANKL and OPG concentrations in patients undergoing orthodontic treatment with clear aligners. The specific objective will be to compare gingival crevicular fluid concentrations of RANKL and OPG among groups according to the application or not of Acceledent® treatment at different time points and frequencies of aligner changes.

DETAILED DESCRIPTION:
Application of intermittent forces by vibration is supposed to be an easy-to-use accelerator of dental movement. The purpose of this study is to determine the effect of intermittent vibrational force application during orthodontic aligner treatment on RANKL and OPG concentrations in crevicular fluid as markers of bone remodelling. This randomized clinical trial will include candidates for malocclusion treatment with aligners, randomly assigned to 3 groups: group A, vibrational forces from onset of treatment; group B, vibrational forces at 6 weeks after treatment onset; and group C, no vibration (controls). The frequency of aligner adjustment will also differ among groups and measurement time points. At different time points, a paper tip will be used to draw crevicular fluid samples from a moving lower incisor for RANKL and OPG analysis using ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of treatment of malocclusion with Invisalign® (Align Technology, San Jose, CAL) using at least 14 sets of aligners
* patients with good general health

Exclusion Criteria:

* smoking habit, poor oral hygiene, the presence of periodontal disease or any other chronic or systemic diseases that could affect bone metabolism or inflammation and the previous or current receipt of medications that could influence bone metabolism (e.g., bisphosphonates).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
RANKL concentration Baseline | Baseline
  Gingival crevicular fluid concentrations of RANKL at baseline
RANKL concentration at 6 weeks | 6 weeks
  Gingival crevicular fluid concentrations of RANKL at 6 weeks
RANKL concentration at 12 weeks | 12 weeks
  Gingival crevicular fluid concentrations of RANKL at 12 weeks
RANKL concentration at 18 weeks | 18 weeks
  Gingival crevicular fluid concentrations of RANKL at 18 weeks
OPG concentration Baseline | Baseline
  Gingival crevicular fluid concentrations of OPG at baseline
OPG concentration at 6 weeks | 6 weeks
  Gingival crevicular fluid concentrations of OPG at 6 weeks
OPG concentration at 12 weeks | 12 weeks
  Gingival crevicular fluid concentrations of OPG at 12 weeks
OPG concentration at 18 weeks | 18 weeks
  Gingival crevicular fluid concentrations of OPG at 18 weeks

SECONDARY OUTCOMES:
Plaque index | Baseline and 18 weeks
  Change in Löe and Silness plaque index scores from baseline to 18 weeks. Values range from 0-3, with higher values indicating more plaque
Gingival index | Baseline and 18 weeks
  Change in Lobenne modified gingival index from baseline to 18 weeks. Values range from 0-3, with higher values indicating more gingival inflammation
Bleeding on probing index | Baseline and 18 weeks
  Change in Bleeding on probing scores from baseline to 18 weeks. Values range from 0-3, with higher values indicating more gingival bleeding
Orthodontic tooth movement achieved | Baseline and 18 weeks
  Amount of tooth movement from baseline to 18 weeks (in mm), measuring tooth displacement from initial to the final position at week 18.

CONTACTS AND LOCATIONS:
Overall Officials: Conchita Martin, Prof, Principal Investigator — Faculty of Odontology, University Complutense Madrid
Locations (1):
- Faculty of Odontology, University Complutense Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teti L, Perez-Idarraga A, Salcedo-Miranda M, Cacho A, Yeste-Ojeda F, Martin C. Randomised Clinical Trial on the Effect of Intermittent Vibrational Force Application During Orthodontic Treatment With Aligners on Root Resorption. Orthod Craniofac Res. 2025 Dec;28(6):1015-1026. doi: 10.1111/ocr.70028. Epub 2025 Sep 10. PMID 40927956